CLINICAL TRIAL: NCT05948384
Title: Comparison of Mirror Therapy and PNF on Lower Extremity Function in Chronic Stroke Patients.
Brief Title: Mirror Therapy Versus PNF on LE Function in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC01540 Shahnoor Syed
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF Group (Active Comparator): For the PNF intervention, we applied a lower extremity hip extension-abduction-internal rotation with knee extension pattern, together with the rhythmic initiation of a repeated stretch and a combination of isotonic techniques. By this we'll target rectus femoris, medial gastrocnemius, lateral gastrocnemius, biceps femoris and semitendinosus musculature of the patient. The session will be given in 2 sets of 5 repetitions with rest of 45 seconds
  Interventions: Other: PNF
- Mirror Therapy Group (Other): Mirror treatment is a sort of motor imagery in which the patient exercises his unaffected limb while looking at himself in the mirror. It involves placing the affected limb behind a mirror. The mirror is positioned so the reflection of the opposing limb appears in place of the hidden limb. The patient then looks into the mirror on the side with unaffected limb and makes "mirror symmetric" movement. It will implemented for about 30 minutes with 2, 2 minutes rest in between. Patient will perform as many repetitions as they could of knee flexion & extension, ankle dorsiflexion & plantarflexion and functional tasks (rolling the foot over the roller, reaching would be accomplished by asking the patient to reach towards objects through his leg e.g. touching the feet to a certain object at a particular height and distance, cycling) depending on patient's ability to do so.
  Interventions: Other: PNF

INTERVENTIONS:
Other: PNF — For the PNF intervention, we applied a lower extremity hip extension-abduction-internal rotation with knee extension pattern, together with the rhythmic initiation of a repeated stretch and a combination of isotonic techniques. By this we'll target rectus femoris, medial gastrocnemius, lateral gastrocnemius, biceps femoris and semitendinosus musculature of the patient. The session will be given in 2 sets of 5 repetitions with rest of 45 seconds

SUMMARY:
Many rehabilitation strategies are being implemented to treat stroke. Constraint-induced movement therapy and robotics are two potentially useful treatment options for rehabilitation. Range of motion exercises, PNF, mirror therapy is also used. Fitness training, high-intensity treatment, and repetitive-task training are all promising strategies that might help improve elements of gait. Repeated task training may also help with transfer functions

DETAILED DESCRIPTION:
PNF and mirror therapy has its effect on chronic stroke patients. Both mirror therapy and PNF work on the concept of neuroplasticity. Neuroplasticity is the ability of the nervous system to change its activity in response to intrinsic or extrinsic stimuli by reorganizing its structure, functions, or connections after injuries. Because of brain plasticity, neurorehabilitation has evolved, as evidenced by numerous physiotherapeutic approaches such as proprioceptive neuromuscular facilitation (PNF) and mirror treatment (MT). The reorganization also includes the expansion of cortical regions, which offer the neural foundation for the recovery or adaption of motor activity following injury.

As the literature supports the individual effects of both techniques in stroke population but as per author's access, there is no literature provide the comparison among both techniques i.e. PNF and mirror therapy in lower limb for chronic stroke patients on gait and functionality. Hence the author established the research question that is there any difference among these techniques in stroke population in terms of its effects and efficiency on gait and functionality. The study will provide an insight to the clinician about which technique has the superior/ better effects for the lower extremity functions in chronic stroke patients thus telling the effects two neurorehabilitation methods i.e. proprioceptive neuromuscular facilitation (PNF) and mirror therapy (MT).

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* ACA stroke
* Ischemic and hemorrhagic stroke
* MMSE grade >24
* Spasticity at modified Ashworth scale between 1 and 2
* Modified Rankin scale 4

Exclusion Criteria:

* Any orthopedic impairment of lower extremity like LLD, fractures, dislocations, amputations, deformity of joint
* Any other neurological condition (multiple sclerosis, Parkinson disease, SCI)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Lower extremity functional scale | 8 week
  a reliable patient-rated outcome measure for assessing lower extremity function. This is a 20-item self-report questionnaire. The highest attainable score is 80 points, signifying excellent function. The lowest possible score is 0, indicating very poor function. It has an outstanding internal reliability (=0.96) and a valid tool. It will be measured at baseline, 4th and 8th week

SECONDARY OUTCOMES:
Dynamic gait index | 8 week
  It assesses the participant's ability to maintain walking balance while reacting to varied task demands under diverse dynamic settings. It is a beneficial test for those who have vestibular and balance issues, as well as those who are at danger of falling. It will be measured at baseline, 4th and 8th week
Time Up and Go Test | 8 week
  Time up and go test is a quick and widely used clinical performance-based measure of lower extremity function, mobility and fall risk with a specificity of 0.70 and sensitivity of 0.57 and reliability of 0.98.The higher the score reflects the worst functional status. It will be measured at baseline, 4th and 8th week
Stroke Specific Quality of Life Scale | 8 week
  It is a patient-centered outcome measure designed to assess health-related quality of life in stroke patients. Patients must answer each question with a reference to the previous week. It is a self-report measure with 49 items divided into 12 areas. A 5-point Likert scale is used to rate the items. The Cronbach alpha ranged from 0.75-0.89. It will be measured at baseline, 4th and 8th week

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Women Institute of Rehabilitation Sciences, Abbottābād, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amarenco P. Transient Ischemic Attack. N Engl J Med. 2020 May 14;382(20):1933-1941. doi: 10.1056/NEJMcp1908837. No abstract available. PMID 32402163
- [Background] Sherin A, Ul-Haq Z, Fazid S, Shah BH, Khattak MI, Nabi F. Prevalence of stroke in Pakistan: Findings from Khyber Pakhtunkhwa integrated population health survey (KP-IPHS) 2016-17. Pak J Med Sci. 2020 Nov-Dec;36(7):1435-1440. doi: 10.12669/pjms.36.7.2824. PMID 33235553
- [Background] Guiu-Tula FX, Cabanas-Valdes R, Sitja-Rabert M, Urrutia G, Gomara-Toldra N. The Efficacy of the proprioceptive neuromuscular facilitation (PNF) approach in stroke rehabilitation to improve basic activities of daily living and quality of life: a systematic review and meta-analysis protocol. BMJ Open. 2017 Dec 12;7(12):e016739. doi: 10.1136/bmjopen-2017-016739. PMID 29233831
- [Background] Gandhi DB, Sterba A, Khatter H, Pandian JD. Mirror Therapy in Stroke Rehabilitation: Current Perspectives. Ther Clin Risk Manag. 2020 Feb 7;16:75-85. doi: 10.2147/TCRM.S206883. eCollection 2020. PMID 32103968